CLINICAL TRIAL: NCT01941355
Title: SheppHeartCABG Shaping Outcomes by Exercise Training and Psycho-education in Phase 1 for Coronary Artery Bypass Grafting Patients
Brief Title: Trial of Rehabilitation in Phase 1 After Coronary Artery Bypass Grafting
Acronym: SheppHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, RN, PhD, Post doc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: SheppHeartCABG
Record Dates: First submitted 2013-09-06; First posted 2013-09-13 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Ischaemic Heart Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Exercise training, psycho-educative (Experimental)
  Interventions: Behavioral: Exercise training component; Behavioral: Psycho-educative component
- Psycho-educative component (Experimental)
  Interventions: Behavioral: Psycho-educative component
- Exercise training component (Experimental)
  Interventions: Behavioral: Exercise training component
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Exercise training component — The physical exercises consist of; deep breathing exercises and breathing exercises using incentive spirometry with expiratory positive pressure airway, cycling exercises during hospitalisation and an individualised exercise programme running from discharge to 4 weeks following surgery.
  Arms: Exercise training component; Exercise training, psycho-educative
Behavioral: Psycho-educative component — The psycho-educative rehabilitation programme consists of four psycho-educative consultations with a specially trained nurse. The last consultation will take place 4 weeks following surgery.
  Arms: Exercise training, psycho-educative; Psycho-educative component

SUMMARY:
Patients undergoing coronary artery bypass graft surgery often experience a range of problems and symptoms related to the procedure and the underlying heart disease. These problems include anxiety and depressive symptoms, immobility issues, complications such as wound seeping, neck and shoulder pains, interrupted and insufficient sleep. Over the last 2 decades, cardiac rehabilitation has become recognized as a significant component in the continuum of care for persons with cardiovascular disease. Furthermore, cardiac rehabilitation has undergone a significant evolution moving from a focused exercise intervention to a comprehensive disease management program. In Guidelines for Coronary Artery Bypass Graft Surgery cardiac rehabilitation is described to include early ambulation during hospitalisation, and outpatient prescriptive exercise training beginning 6-8 weeks following surgery. Our hypothesis is that physical exercise with moderate intensity and a psycho-educative component as a part of cardiac rehabilitation can begin in early postoperatively during hospitalising. Results from studies on phase 1 rehabilitation in coronary artery bypass graft surgery patients are promising. However, no randomised trials have been conducted, and evidence is therefore lacking.

The objective of this pilot trial is to investigate the effect of a phase 1 comprehensive cardiac rehabilitation programme consisting of a psycho-educative component, an exercise-training component including pulmonary training, cycling, neck and shoulder exercises, these in combination plus treatment as usual and treatment as usual in patients who undergo coronary artery bypass grafting.

SheppHeartCABG is an investigator-initiated 2 x 2 factorial randomised clinical pilot trial with blinded outcome assessment. Recruitment from one site with 1:1:1:1 central randomisation to phase 1 rehabilitation; 1) exercise-training plus usual care, 2) psycho-educative plus usual care 3) exercise-training and psycho-educative plus usual, 4) usual care alone.

DETAILED DESCRIPTION:
The explorative outcome measures consist of two parts: physical capacity and mental and physical health. Physical capacity is measured by peak VO2 max and 6 minutes' walk test at discharge and 4 weeks following surgery. Perceived mental and physical health is measured by the Medical Outcome Study Short Form 36 (SF-36) at admission, discharge and 4 weeks following surgery. Furthermore questionnaires measuring anxiety and depression (Hospital Anxiety and Depression Scale), health-related quality of life (HeartQoL), fatigue (MFI-20) cognitive and emotional representation of illness (B-IPQ), physical activity (IPAQ), self-rated health (EQ-5D), sleep (PSQI) and pain (ÖMPSQ)

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Persons with ischaemic heart disease referred to elective coronary artery bypass graft surgery.
* Speaks and understands Danish.
* Provide written informed consent.

Exclusion Criteria:

* Patients at intermediate or high risk according to their cardiovascular status
* Patients with illness limiting the ability to exercise.
* Patients without permanent residence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen uptake (VO2) between groups | At hospital discharge and 4 weeks following surgery
Change in self-reported health measured by SF-36 between groups | At hospital discharge and 4 weeks following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Selina K Berg, PhD, Post doc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark